CLINICAL TRIAL: NCT05366855
Title: A Phase 3, Long-Term Extension Study to Evaluate the Safety and Efficacy of Imsidolimab (ANB019) in the Treatment of Adult Subjects With Generalized Pustular Psoriasis
Brief Title: Long-Term Safety and Efficacy of Imsidolimab (ANB019) in Subjects With Generalized Pustular Psoriasis
Acronym: GEMINI-2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: AnaptysBio has concluded the GEMINI-2 trial, with all trial participants having been treated with imsidolimab for approximately six months and the furthest patient having been treated through 92 weeks
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANB019-302
Record Dates: First submitted 2022-04-25; First posted 2022-05-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2024-08

CONDITIONS: Generalized Pustular Psoriasis
Keywords: IL-36 receptor; Interluekin 36; Imsidolimab
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- IV +SC Imsidolimab (Active Comparator): IV loading dose followed by subcutaneous Imsidolimab
  Interventions: Biological: Imsidolimab
- SC Imsidolimab (Active Comparator): Subcutaneous Imsidolimab
  Interventions: Biological: Imsidolimab
- SC Placebo (Placebo Comparator): Subcutaneous Placebo
  Interventions: Other: Placebo
- Standard of Care (No Intervention): Any available therapy

INTERVENTIONS:
Biological: Imsidolimab — Solution for infusion; Solution for injection
  Other Names: ANB019
  Arms: IV +SC Imsidolimab; SC Imsidolimab
Other: Placebo — Solution for injection
  Arms: SC Placebo

SUMMARY:
This is a Phase 3, long term extension study to evaluate the safety and efficacy of imsidolimab compared with placebo in adult subjects with generalized pustular psoriasis (GPP).

DETAILED DESCRIPTION:
This study will also evaluate the pharmacokinetic (PK) profile of imsidolimab and explore the immunogenicity of imsidolimab in subjects with GPP

ELIGIBILITY:
Inclusion Criteria:

* Subject participated in the preceding placebo-controlled Phase 3 study ANB019-301 and completed at least the Week 1 visit of the ANB019-301 study without the use of rescue/prohibited medication for GPP
* Subject must be a candidate for prolonged GPP treatment according to the Investigator's judgment

Exclusion Criteria:

* Use of prohibited medications between the last visit of the ANB019-301 study and the Day 1 visit of the ANB019-302 study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2024-07-17 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Week 24
  Incidence of adverse events

CONTACTS AND LOCATIONS:
Locations (67):
- United States (6):
  - Site 109, Largo, Florida
  - Site 105, Louisville, Kentucky
  - Site 10-101, Ann Arbor, Michigan
  - Site 101, Ann Arbor, Michigan
  - Site 108, Dallas, Texas
  - Site 102, Springville, Utah
- Australia (2):
  - Site 35-101, Melbourne
  - Site 35102, Sydney
- France (2):
  - Site 16-102, Nantes
  - Site 16-101, Paris
- Georgia (5):
  - Site 59104, Batumi
  - Site 59-101, Tbilisi
  - Site 59-105, Tbilisi
  - Site 59102, Tbilisi
  - Site 59103, Tbilisi
- Germany (4):
  - Site 17102, Bensheim
  - Site 17104, Bonn
  - Site 17103, Hanau
  - Site 17105, Würzburg
- Malaysia (10):
  - Site 42104, Cheras
  - Site 42-107, Johor Bahru
  - Site 42106, Johor Bahru
  - Site 42105, Kota Bharu
  - Site 42-110, Kuala Lumpur
  - Site 42101, Kuala Lumpur
  - Site 42102, Muar town
  - Site 42-108, Pulau Pinang
  - Site 42103, Putrajaya
  - Site 42-109, Selayang Baru Utara
- Morocco (3):
  - Site 64-102, Casablanca
  - Site 64-103, Casablanca
  - Site 64-101, Oujda
- Poland (5):
  - Site 30104, Krakow
  - Site 30105, Lodz
  - Site 30103, Ossy
  - Site 30101, Rzeszów
  - Site 30102, Wroclaw
- Romania (3):
  - Site 31-102, Bucharest
  - Site 31-101, Cluj-Napoca
  - Site 31-103, Iași
- South Korea (4):
  - Site 45101, Pusan
  - Site 45102, Seoul
  - Site 45103, Seoul
  - Site 45104, Seoul
- Spain (5):
  - Site 24-101, Barcelona
  - Site 24-104, Las Palmas de Gran Canaria
  - Site 24-102, Madrid
  - Site 24-103, Madrid
  - Site 24-105, Valencia
- Taiwan (4):
  - Site 63101, Kaohsiung City
  - Site 63102, Taipei
  - Site 63103, Taipei
  - Site 64104, Taipei
- Thailand (4):
  - Site 46101, Bangkok
  - Site 46102, Chiang Mai
  - Site 46104, Khon Kaen
  - Site 46103, Pathum Thani
- Tunisia (3):
  - Site 62-101, Sfax
  - Site 62-102, Sousse
  - Site 62-103, Tunis
- Turkey (Türkiye) (7):
  - Site 33-101, Ankara
  - Site 33-103, Antalya
  - Site 33-105, Istanbul
  - Site 33-106, Istanbul
  - Site 33-107, Istanbul
  - Site 33-102, Kayseri
  - Site 33-104, Nilufer

IPD SHARING:
Plan to Share IPD: No